CLINICAL TRIAL: NCT03972085
Title: Comparison of Conservative Treatment With and Without Neural Gliding Exercise for Patients With Low Back Pain
Brief Title: Neural Gliding Exercise for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Vedat KURT, Principal investigator, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80558721/153-002
Record Dates: First submitted 2019-05-28; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Neurodynamics
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patient received neural gliding exercises in addition electrotehrapy sessions.
  Interventions: Other: Neural gliding exercises; Other: Electrotherapy sessions
- Group 2 (Active Comparator): Patient received only electrotherapy sessions
  Interventions: Other: Electrotherapy sessions

INTERVENTIONS:
Other: Neural gliding exercises — Neural gliding exercises: In addition to the Electrotherapy procedure, patients were asked to actively perform knee extension, ankle dorsiflexion and head extension in the slumped posture followed by simultaneous ankle plantar flexion together with knee and head flexion (10 repetitions in 1 minute). Patients performed the exercises under a home-based program for 5 days of the week during a total period of 3 weeks.
  Electrotherapy sessions: Local Hot Pack (30 minutes), Chattanoga™ TENS (20 minutes, 80-180 Hz frequency, 50-100 wavelength) and Chattanoga™ ultrasound (1 Mhz frequency, 3 W/cm2 3 minutes) were applied for 5 days per week during a total period of 3 weeks. Subjects in ETG did not do any other exercise approach.
  Other Names: Electrotherapy sessions
  Arms: Group 1
Other: Electrotherapy sessions — Electrotherapy sessions: Local Hot Pack (30 minutes), Chattanoga™ TENS (20 minutes, 80-180 Hz frequency, 50-100 wavelength) and Chattanoga™ ultrasound (1 Mhz frequency, 3 W/cm2 3 minutes) were applied for 5 days per week during a total period of 3 weeks. Subjects in ETG did not do any other exercise approach.

SUMMARY:
Low back pain is a very common problem that causes pain, disability, gait and balance problems. Neurodynamic techniques is used for treatment of low back pain. The aim of the study is comparing the effects of electrotherapy and neural mobilization techniques on pain, functionality, gait and balance.

DETAILED DESCRIPTION:
There are many physiotherapy modalities in the treatment of low back pain (LBP). Electrotherapy procedures, manual therapy techniques, kinesiotherapy and specific exercises are among those that are frequently used. In neural mobilization techniques, which began to gain popularity in 1990s, neural tissue and the surrounding structures are glided or tensioned to mobilize them. Neural mobilization is thought to have a positive effect on symptoms by inducing intraneural circulation, axoplasmic flow, and neural visco-elasticity and sensitivity associated with the connective tissue. There are studies in which this modality has yielded therapeutic success in terms of both pain and functionality, particularly in lumbar region and lower limb disorders where neural mechanosensitivity is increased.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scoring below 70 degrees in the straight leg raise test
* received no physiotherapy until at least 6 months before initial evaluation

Exclusion Criteria:

* subjects who were unable to walk independently,
* who had systemic diseases besides LBP,
* who underwent spinal and lower limb surgery,
* who scored above 70 degrees in the straight leg raise test,
* used analgesics within 48 hours before initial evaluation were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-11-07 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for pain levels | 3 weeks
  The VAS was used to assess the participants' pain levels. In the VAS, patients are asked to mark the severity of their pain on a scale from 0 to 10. The VAS ranges from '0' representing no pain and '10' representing the worst pain.

SECONDARY OUTCOMES:
Oswestry Disability Index | 3 weeks
  The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University, Kütahya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No